CLINICAL TRIAL: NCT00922987
Title: Non-Interventional Study (NIS) With Lyrica In Patients With Epilepsy As Adjunctive Therapy Of Partial Seizures To Reduce Seizure Frequency
Brief Title: Clinical Study With Lyrica In Patients Suffering From Epilepsy
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081236
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2011-07

CONDITIONS: Neuralgia; Epilepsy
Keywords: lyrica pregabalin epilepsy partial seizures
MeSH Terms: conditions — Neuralgia; Epilepsy | interventions — Pregabalin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lyrica: Adult patients with partial seizures (type of epilepsy). Inclusion criteria according to Summary of Product Characteristics
  Interventions: Drug: Lyrica (pregabalin)

INTERVENTIONS:
Drug: Lyrica (pregabalin) — The daily dose may range from 150mg to 600mg, administered as two single doses. The treatment should be started with 150mg daily dose (2x75mg). Depending on response and tolerability after 7 days may the dose be increased to 300mg/day (2x150mg) and after further 7 days to maximum dose 600mg/day (2x300mg)

SUMMARY:
Clinical study with Lyrica (pregabalin) in patients suffering from epilepsy. This drug is used as adjunctive therapy with one or more antiepileptics. Lyrica has potential to reduce seizure frequency.

DETAILED DESCRIPTION:
- Included all adult patients with partial seizures and without contraindications according to Summary of Product Characteristics (SmPC).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with partial seizures.

Exclusion Criteria:

* Contraindications according to Summary of Product Characteristics (SmPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adult patiens with partial seizures.
  * Other inclusion criteria according to Summary of Product Characteristics (SmPC).
Sampling Method: Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- Slovakia (44):
  - Pfizer Investigational Site, Banská Bystrica
  - Pfizer Investigational Site, Bardejov
  - Pfizer Investigational Site, Bojnice
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Čadca
  - Pfizer Investigational Site, Dolný Kubín
  - Pfizer Investigational Site, Dubnica nad Váhom
  - Pfizer Investigational Site, Dunajská Streda
  - Pfizer Investigational Site, Handlová
  - Pfizer Investigational Site, Hlohovec
  - Pfizer Investigational Site, Humenné
  - Pfizer Investigational Site, Kemarok
  - Pfizer Investigational Site, Komárno
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Krompachy
  - Pfizer Investigational Site, Levice
  - Pfizer Investigational Site, Levoča
  - Pfizer Investigational Site, Liptovský Mikuláš
  - Pfizer Investigational Site, Malacky
  - Pfizer Investigational Site, Martin
  - Pfizer Investigational Site, Modra
  - Pfizer Investigational Site, Myjava
  - Pfizer Investigational Site, Nitra
  - Pfizer Investigational Site, Nové Mesto nad Váhom
  - Pfizer Investigational Site, Nové Zámky
  - Pfizer Investigational Site, Piešťany
  - Pfizer Investigational Site, Poltár
  - Pfizer Investigational Site, Prešov
  - Pfizer Investigational Site, Púchov
  - Pfizer Investigational Site, Ružomberok
  - Pfizer Investigational Site, Sereď
  - Pfizer Investigational Site, Skalica
  - Pfizer Investigational Site, Snina
  - Pfizer Investigational Site, Spišská Nová Ves
  - Pfizer Investigational Site, Šahy
  - Pfizer Investigational Site, Šurany
  - Pfizer Investigational Site, Trebišov
  - Pfizer Investigational Site, Trenčín
  - Pfizer Investigational Site, Trnava
  - Pfizer Investigational Site, Trstená
  - Pfizer Investigational Site, Vranov Nad Toplov
  - Pfizer Investigational Site, Zlaté Moravce
  - Pfizer Investigational Site, Zvolen
  - Pfizer Investigational Site, Žilina

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081236&StudyName=Clinical%20Study%20With%20Lyrica%20In%20Patients%20Suffering%20From%20Epilepsy

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 286 participants were assigned to treatment. At 1 of study sites, lack of archival of study files, source documentation, missing informed consent forms and large data discrepancies led to exclusion of all data from this site (N=5), as data could not be verified. Removal of these 5 participants did not change interpretation of results.
Groups:
- Pregabalin: Pregabalin (Lyrica) at a dose ranging from 150 milligrams (mg) to 600 mg administered as two single doses, daily until Week 16.
Period: Overall Study
Arm/Group | Pregabalin
Started | 281
Completed | 277
Not Completed | 4
Not completed — Insufficient clinical response | 1
Not completed — Protocol Violation | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (13.7)
Sex/Gender, Customized [Number; unit: participants]
  Male | 137
  Female | 142
  Unspecified | 2
Comorbidities in the past [Number; unit: Participants]
  Hypercoagulation | 1
  Transposition of great vessels | 1
  Hypothyroidism | 1
  Dyspepsia | 1
  Gastric ulcer | 1
  Ill-defined disorder | 4
  Pyrexia | 1
  Hepatitis toxic | 1
  Hepatitis non-A non-B | 1
  Herpes zoster | 1
  Meningitis | 1
  Brain contusion | 4
  Concussion | 2
  Extradural haematoma | 1
  Femur fracture | 1
  Head injury | 2
  Subdural haematoma | 1
  Traumatic brain injury | 5
  Hepatitis B surface antigen positive | 1
  Back pain | 1
  Muscle spasms | 1
  Brain neoplasm | 2
  Meningioma | 5
  Pleura carcinoma | 1
  Central nervous system lesion | 1
  Cerebral hemorrhage | 1
  Cerebrovascular accident | 3
  Convulsion | 1
  Demyelination | 1
  Encephalitis | 3
  Encephalomalacia | 1
  Encephalopathy | 3
  Epilepsy | 1
  Headache | 1
  Hypotonia | 1
  Hypoxic encephalopathy | 1
  Neuritis | 1
  Delivery | 1
  Alcohol abuse | 1
  Depression | 2
  Psychotic disorder | 1
  Neonatal asphyxia | 1
  Pulmonary embolism | 1
  Appendicectomy | 1
  Cholecystectomy | 1
  Craniotomy | 1
  Glaucoma surgery | 1
  Hysterectomy | 1
  Inguinal hernia repair | 1
  Meningioma surgery | 1
  Spinal anaesthesia | 1
  Spinal laminectomy | 1
  Strabismus correction | 1
  Subdural haematoma evacuation | 1
  Hypertension | 2
Prior anti-epileptic medications [Number; unit: Participants]
  Carbamazepine | 135
  Cinolazepam | 1
  Clonazepam | 7
  Ergenyl chrono | 27
  Gabapentin | 2
  Lacosamide | 4
  Lamotrigine | 57
  Levetiracetam | 30
  Oxcarbazepine | 12
  Phenobarbital | 2
  Phenytoin | 14
  Pregabalin | 15
  Primidone | 1
  Sultiame | 1
  Topiramate | 40
  Valproate sodium | 24
  Valproic acid | 66
  Vigabatrin | 1
  Zentronal | 1
28-Day partial seizure frequency [Mean (Standard Deviation); unit: seizures] — The partial seizure frequency for the baseline period was the total number of partial seizures recorded for that period at Visit 0 (week 0). This was evaluated for 264 participants.
  seizures | 2.31 (1.33)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a 50 Percent or Greater Reduction From Baseline in 28 Day Partial Seizure Frequency
Description: Responder rate was defined as the percentage of participants with at least a 50% reduction in 28-day partial seizure frequency from baseline during the maintenance phase (Week 4 - Week 16). The percent change in partial seizure frequency in the maintenance phase was the change from baseline in partial seizure frequency * 100, divided by the partial seizure frequency at the baseline visit.
Time Frame: Baseline through week 16 or early termination (ET)
Population: The modified full analysis set (MFAS) included all participants who received at least 1 dose of the study drug and who had at least one baseline seizure. Participants who discontinued during first 4 weeks titration phase were regarded as missing and were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 260
Percentage of participants | 85.00 [80.66 to 89.34]

2. Secondary Outcome: Percentage Change From Baseline in 28 Day Partial Seizure Frequency at Final Visit
Description: The partial seizure frequency for the baseline period was the total number of partial seizures recorded for that period at Visit 0 (week 0). For each participant's final visit, the 28 day partial seizure frequency equals total number of partial seizures since the last visit * 28 divided by total number of days since the last visit. For percent change from baseline: change from baseline in partial seizure frequency*100 divided by partial seizure frequency at baseline visit.
Time Frame: Baseline and week 16 or ET
Population: MFAS included all participants who received at least 1 dose of the study drug and who had at least one baseline seizure. Participants who discontinued during first 4 weeks titration phase were regarded as missing and were excluded from the analysis. Analysis was done using last observation carried forward (LOCF) method.
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | Pregabalin
Number analyzed (Participants) | 262
percent change | -100.00 [-100.00 to -87.93]
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < 0.0001, Signed Rank Test

3. Secondary Outcome: Number of Participants With no Seizures (Partial or Other) During the Last 4 Weeks in the Study
Description: Participants were regarded as seizure-free if no seizures (partial or other) were reported for the participant during the last 4 weeks in the study.
Time Frame: Week 4 through week 16 or ET
Population: MFAS: Data collected during the titration phase, i.e. prior to Visit 2 (Week 4) were not analyzed for this endpoint. Only participants who did not discontinue in the first 4 weeks after the baseline visit (titration phase) and had at least 4 weeks of seizure data during the maintenance phase were analyzed for this endpoint.
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 243
Participants | 172

4. Secondary Outcome: Change From Baseline in Visual Analog Scale of Anxiety (VAS-A) Scores at Week 4 and Final Visit
Description: VAS-A consists of a visual analog scale ranging from, 0 mm (no anxiety) to 100 mm (extreme anxiety).
Time Frame: Baseline, week 4 and week 16 or ET
Population: Full Analysis Set (FAS): Included all participants who received at least 1 dose of study drug. Participants who did not have the minimum required data for the statistical summary were treated as missing. Analysis was done using LOCF method.
Measure: Mean (95% Confidence Interval); unit: millimeter (mm)
Arm/Group | Pregabalin
Number analyzed (Participants) | 279
millimeter (mm)
  Baseline | 54.12 [51.32 to 56.92]
  Change at Week 4 | -13.60 [-15.37 to -11.84]
  Change at Week 16 or ET | -26.16 [-28.73 to -23.59]

5. Secondary Outcome: Number of Participants With Categorical Scores on Clinical Global Impression of Severity (CGI-S)
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected.
Time Frame: Baseline
Population: FAS: Included all participants who received at least 1 dose of study drug. Participants who did not have the minimum required data for the statistical summary were treated as missing.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 269
participants
  Not Assessed | 0
  Normal, not at all ill | 17
  Borderline ill | 25
  Mildly ill | 64
  Moderately ill | 118
  Markedly ill | 32
  Severely ill | 8
  Among the most extremely ill participants | 5

6. Secondary Outcome: Number of Participants With Change in Clinical Global Impression of Severity (CGI-C) From Baseline at Final Visit
Description: The CGI-C scale measures a physician's global impression of a participant's clinical condition at final visit in terms of change relative to the start of treatment (CGI-C).
  At final visit, the participants CGI-C will be categorized into a three point scale as: improvement: CGI response of very much improved, much improved or minimally improved; no change: CGI response of no change; worsening: CGI response of very much worse, much worse or minimally worse.
Time Frame: Week 16 or ET
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 273
Participants
  Not Assessed | 0
  Very much improved | 48
  Much improved | 145
  Minimally improved | 50
  No change | 29
  Minimally worse | 0
  Much worse | 1
  Very much worse | 0

7. Secondary Outcome: Change From Baseline in Medical Outcome Study (MOS) Sleep Scale Sub-scores at Week 16 or ET
Description: MOS: participant rated questionnaire, assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); 7 subscales rated 1 (all the time) to 6 (none of the time): sleep disturbance, snoring, awaken short of breath (SOB) or with a headache, somnolence adequacy, and sleep quantity. Transformed scores (actual raw score minus lowest possible score divided by possible raw score range multiplied by 100); sub-scales total score range= 0-100; higher score indicates greater intensity of attribute.
Time Frame: Baseline and week 16 or ET
Population: The FAS included all participants who received at least 1 dose of the study drug and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 281
Units on a scale
  Baseline: Sleep Problems Index I | 44.72 (18.61)
  Baseline: Sleep Problems Index II | 44.55 (18.59)
  Baseline: Sleep Disturbance | 44.31 (22.44)
  Baseline: Snoring | 33.71 (26.19)
  Baseline: Awaken Short of Breath | 34.41 (26.45)
  Baseline: Quantity of Sleep (hours) | 6.77 (1.23)
  Baseline: Sleep Adequacy | 45.50 (22.12)
  Baseline: Somnolence | 37.19 (20.58)
  Change at Week 16: Sleep Problems Index I | -16.93 (18.52)
  Change at Week 16: Sleep Problems Index II | -19.44 (17.27)
  Change at Week 16: Sleep Disturbance | -25.04 (19.49)
  Change at Week 16: Snoring | -10.14 (18.88)
  Change at Week 16: Awaken Short of Breath | -16.55 (24.26)
  Change at Week 16: Quantity of Sleep (hours) | 0.92 (1.02)
  Change at Week 16: Sleep Adequacy | 9.27 (29.76)
  Change at Week 16: Somnolence | -17.72 (16.45)

8. Other Pre Specified Outcome: Number of Participants With Concomitant Drug Treatments
Description: Concomitant drug (any drug other than, and in addition to, the study drug) taken for any period of time during the study.
Time Frame: Baseline through Week 16 or ET
Population: Safety analysis set included all enrolled participants who received 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 281
participants
  Acetylsalicylic acid | 8
  All other therapeutic products | 1
  Allopurinol | 1
  Alprazolam | 4
  Aminophylline | 1
  Amlodipine | 3
  Amlodipine Besilate | 1
  Asasantin | 2
  Atenolol | 1
  Atorvastatin | 2
  Baclofen | 1
  Betahistine | 1
  Betahistine hydrochloride | 1
  Betaxolol hydrochloride | 1
  Biselect | 2
  Bisoprolol | 2
  Carbamazepine | 114
  Citalopram | 1
  Clonazepam | 8
  Clopidogrel | 2
  Clopidogrel sulfate | 1
  Coversum combi | 1
  Desloratadine | 1
  Diazepam | 2
  Diclofenac | 2
  Digoxin | 1
  Drug unspecified | 4
  Ergenyl chrono | 27
  Escitalopram | 3
  Fenofibrate | 1
  Fentanyl | 1
  Fluphenazine decanoate | 1
  Folic acid | 1
  Furosemide | 1
  Gabapentin | 2
  Gingko biloba | 1
  Gingko biloba extract | 5
  Gliclazide | 1
  Hyzaar | 1
  Ibuprofen | 1
  Imidapril hydrochloride | 1
  Insulin | 3
  Ipratropium bromide | 1
  Lacosamide | 3
  Lamotrigine | 54
  Levetiracetam | 30
  Levothyroxine sodium | 1
  Magnesium | 1
  Metamizole sodium | 1
  Metformin hydrochloride | 2
  Molsidomine | 1
  Oxazepam | 1
  Oxcarbazepine | 11
  Paracetamol | 1
  Pentoxifylline | 1
  Perindopril | 1
  Perindopril arginine | 1
  Phenobarbital | 1
  Phenytoin | 11
  Piracetam | 6
  Pregabalin | 66
  Primidone | 1
  Ramipril | 2
  Seretide mite | 1
  Sertraline | 3
  Silymarin | 1
  Sultiame | 1
  Telmisartan | 1
  Theophylline | 1
  Thioctic acid | 2
  Tianeptine | 1
  Tiapride | 2
  Ticlopidine | 1
  Ticlopidine hydrochloride | 1
  Tocopherol | 2
  Topiramate | 34
  Tramadol | 1
  Trandolapril | 3
  Trazodone hydrochloride | 1
  Valproate sodium | 23
  Valproic acid | 55
  Venlafaxine | 1
  Venlafaxine hydrochloride | 1
  Verapamil hydrochloride | 1
  Vinpocetine | 2
  Warfarin sodium | 1

9. Other Pre Specified Outcome: Number of Participants With Concomitant Co-morbidities
Description: Participants who had a concomitant co-morbidity during the study for any period of time from baseline through to Week 16 (Final Visit); participants with more than one concomitant co-morbidity were counted for each of the co-morbidity classes applicable.
Time Frame: Baseline through week 16 or ET
Population: Safety analysis set included all enrolled participants who received 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 281
participants
  Anaemia | 1
  Thrombocytopenia | 1
  Cardiomyopathy | 1
  Coronary artery disease | 3
  Myocardial ischaemia | 4
  Sturge-Weber syndrome | 1
  Deafness | 1
  Hypoacusis | 1
  Vertigo | 1
  Autoimmune thyroiditis | 1
  Endocrine disorder | 1
  Goitre | 1
  Hypothyroidism | 1
  Reflux oesophagitis | 1
  Hepatic fibrosis | 1
  Liver disorder | 4
  Multiple allergies | 1
  Seasonal allergy | 1
  Neuroborreliosis | 1
  Injury | 1
  Diabetes mellitus | 6
  Hyperlipidemia | 2
  Obesity | 1
  Type 1 diabetes mellitus | 1
  Type 2 diabetes mellitus | 1
  Mucoskeletal pain | 1
  Osteoarthritis | 3
  Osteoporosis | 2
  Spinal disorder | 2
  Brain neoplasm malignant | 1
  Oligodendroglioma | 1
  Cerebral ischaemia | 2
  Cerebrovascular accident | 1
  Dementia Alzheimer's type | 1
  Dizziness | 1
  Encephalopathy | 1
  Grand mal convulsion | 1
  Headache | 1
  Hemiparesis | 1
  Mental retardation | 3
  Migraine | 1
  Migraine without aura | 1
  Neuropathy peripheral | 1
  Polyneuropathy | 1
  Anxiety | 6
  Anxiety disorder | 1
  Depression | 11
  Generalised anxiety disorder | 1
  Post-traumatic stress disorder | 1
  Psychotic disorder due to medical condition | 4
  Schizophrenia | 2
  Diabetic neuropathy | 1
  Nephropathy | 1
  Asthma | 1
  Chronic obstructive pulmonary disease | 2
  Hypertension | 28
  Post thrombotic syndrome | 1

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 1/281
Other Adverse Events (participants affected / at risk) | 4/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=281)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=281)
Weight increased (Investigations) | 4 (4)
Somnolence (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
On review of blinded data it was decided that an additional analysis set, MFAS was required. MFAS was created for analysis of seizure data. The outcomes related to seizure data were therefore analyzed for MFAS population and not FAS population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.